CLINICAL TRIAL: NCT00144716
Title: Clinical Evaluation of Combined Use of ITN's and Plant-based Insect Repellent Against Malaria in the Amazon
Brief Title: Evaluation of Combined Use of ITN's and Insect Repellents Against Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ITDCVG30
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: Vector Control; repellent; ITN's; malaria; Amazon
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Device: Insect Repellent plus Insecticide Treated Net

SUMMARY:
Insecticide Treated Nets (ITN's) offer good protection against malaria in Africa where the vector mosquitoes feed indoors late at night. However, in other parts of the world like South America, vectors feed earlier in the evening before people go to bed. In such cases it may be necessary to use alternative treatments in the evening to supplement the efficacy of ITN's. This study compares 2 matched groups of households in the Bolivian Amazon. One group will be given ITN's plus a plant-based insect repellent in the evening, the other has ITN's plus a placebo lotion. Households are monitored over a full malaria season to record numbers of malaria cases.

DETAILED DESCRIPTION:
There is little doubt that the use of insecticide treated bed nets (ITN's) is one of the most successful means of reducing malaria in Africa. However, vectors in this region tend to be late night, indoor feeders. Vector species in other parts of the world may not be so susceptible to this form of vector control. In much of Central & Southern America, the major vectors such as An. darlingi and An. albitarsis have a feeding peak between 8 - 10pm, before most people retire to bed. Similarly, the major vector in much of S.E. Asia, An. dirus, seldom enters homes to feed. In these circumstances it is unlikely ITN's alone will provide adequate protection. Supplemental use of skin applied insect repellents may be an effective method of personal protection in the hours between dusk and retiring to bed. It would also prove useful for those individuals working late or moving early into the forest where exophagic species are encountered. As yet, there have been no robust clinical evaluations of combined ITN and repellent use. This double blind, placebo-controlled study is designed to evaluate the efficacy of combined ITN and plant based insect repellent use to reduce P. falciparum in the Bolivian Amazon in a region where ITN's alone are likely to be ineffective.

The study is a double-blind, placebo-controlled clinical evaluation. 1000 households will be used and 5 individuals age 10 + will be entered into the study from each. Recruitment will cover all rural communities in Vaca Diez and Pando Provinces, Department of Beni in the Bolivian Amazon Region, plus the outer 10 % of periurban districts of the 2 major towns in the region, Riberalta and Guayaramerin. A maximum of 20 % of households in any one location will be used, thus avoiding any effect of diversion of insects from treatment to placebo homes. Likewise, each house used will be a minimum of 25m from any other in the study. Baseline surveys will be conducted on each individual and informed written consent will be collected. Treatment (30 % L.E.) / placebo (0.1 % clove oil in alcohol) marked A or B will be allocated (50:50) at random, and all individuals in both groups will be provided with an ITN. Compliance questionnaires, collection of old bottles and distribution of fresh bottles will be conducted every 4 weeks. Everyone will receive personal instruction on how to apply repellent to arms & legs each evening at dusk and left a pictorial instruction sheet on how to measure 10 ml using the bottle lid. Compliance threshold will be set at 10% and monitored by measuring any residual product on collection and recording of nightly use. A more realistic measure of compliance will be gained through occasional evening spot checks of households by the local health workers. Finger prick blood samples will be collected at baseline and monthly throughout the study by trained & approved field staff. P. falciparum infection will be diagnosed by Paracheck® dipstick test, thus overcoming problems of recrudescence of P. vivax. Positive cases will be referred to the local health centre for treatment. The timing of the visits means the majority of malaria episodes will be detected as the Paracheck® test can detect antibodies in blood for around 3 weeks post treatment. In addition to the use of our monthly questionnaires, any episodes missed are highly likely to be recorded, as we are employing the same local health workers in each area, and blood slides are routinely taken at the local health centres. Outcome determination will constitute a series of monthly cross-sectional prevalence surveys, and, as positive cases are treated, this is equivalent to a measure of average prevalence of infection for each house.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Available for 4 x monthly follow ups.
* 5 or more individuals in household.

Exclusion Criteria:

* Allergy to repellents / plants.
* Malaria positive at baseline.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4250
Dates: Start 2003-06; Study Completion 2003-10

PRIMARY OUTCOMES:
Reduction in cases of malaria

SECONDARY OUTCOMES:
Reduction in all-cause fevers

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Hill, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine

REFERENCES:
- [Derived] Hill N, Lenglet A, Arnez AM, Carneiro I. Plant based insect repellent and insecticide treated bed nets to protect against malaria in areas of early evening biting vectors: double blind randomised placebo controlled clinical trial in the Bolivian Amazon. BMJ. 2007 Nov 17;335(7628):1023. doi: 10.1136/bmj.39356.574641.55. Epub 2007 Oct 16. PMID 17940319